CLINICAL TRIAL: NCT06455163
Title: Eerder Erbij: Een Vroege Ondersteuning Voor Mensen Met Dementie en Hun Mantelzorgers. The Path Towards Offering Timely Support for People With Dementia and Their Caregivers
Brief Title: Eerder Erbij: The Path Towards Offering Timely Support for People With Dementia and Their Caregivers
Acronym: EE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Sanne Balvert, Principal Investigator, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 852002106
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Dementia, Mild
Keywords: Early-stage dementia; Informal caregiver; Informal care
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eerder Erbij (intervention group) (Experimental): Informal caregivers and people with dementia assigned to the intervention group will receive the 6-week intervention "Eerder Erbij".
  Interventions: Other: Eerder Erbij
- Usual/standard care (control group) (No Intervention): Participants in the comparison condition will continue to receive usual care. Care for people with dementia in the Netherlands varies across municipalities, but the majority lives at home and especially earlier stages of the disease, most people living with dementia and their informal caregivers use no or very little formal care, apart from occasional visitors to GP or by case manager.
  The control group will be shared with another collaborating study from 'Maastricht University', which has the same goals, applies the same inclusion criteria, applies the same study procedures, and obtains the same outcomes. This implies that the data of the participants recruited for the control group for this study will be shared with the collaborating study.

INTERVENTIONS:
Other: Eerder Erbij — The intervention (Eerder Erbij, EE) is a person-centred, manual-based intervention consisting of education, information and a support group for persons in the early stage of dementia and their main informal caregiver (e.g. spouse, relative), who receive little or no formal care. The intervention will discuss the effects of dementia, and how to cope and adjust to those effects. It will take place in small group sessions led by a health care professional (e.g. casemanager) and is intended for both the person with dementia and the caregiver. The intervention will be personalised to meet needs, interests and strengths of the dyad by discussing the sessions content at the start of the intervention.
  Arms: Eerder Erbij (intervention group)

SUMMARY:
INTRODUCTION AND RATIONALE

It has been estimated that at least 50% of the home living persons with dementia in the Netherlands receive little or no formal care and support (Zorgstandaard Dementie, 2013). Reasons why persons with dementia and their informal caregivers receive no formal care vary, include absence of diagnosis, denial of illness, embarrassment or the complexity of the care and referral system. A common concern among health care professionals is that by the time the person with dementia or informal caregiver do seek or receive formal care it may be too late. The difficulties at home may already be so severe that there is little that community-based care can do and admission to residential care may follow soon after. Appropriate support at an earlier stage may prevent more serious difficulties and postpone admission to residential care. Therefore, health care professionals are looking for strategies to reach persons with dementia and caregivers in an earlier stage of dementia and encourage them to accept some form of help or support. The rationale of this study is to investigate how persons living with dementia and their close others can be encouraged to accept support and whether support at an early stage is effective in preventing severe deterioration in wellbeing, behavioural difficulties and high care costs later on.

OBJECTIVES

* Estimate the effect of EE on caregiver self-efficacy compared to usual care
* Estimate the effect of EE on the total care costs of caregiver and person with dementia compared to usual care
* Estimate the cost-effectiveness and cost-utility of EE compared to usual care
* Perform a process evaluation to monitor delivery of EE and experiences of persons with dementia, caregivers and care professionals
* Explore treatment responsiveness of EE in terms of self-efficacy and quality of life

STUDY DESIGN

Pragmatic, cluster randomised controlled trial.

STUDY POPULATION

Informal caregivers and people with early-stage dementia, who are community dwelling and receive little or no dementia-related formal ADL care.

INTERVENTION

The intervention (Eerder Erbij, EE) is a person-centred, manual-based intervention consisting of education, information and a support group.

MAIN STUDY PARAMETERS/ENDPOINTS

Primary: self-efficacy. Cost-utility: EQ5D, RUD. Secondary: quality-of-life, caregiver burden.

DATA COLLECTION

Measurements consist of questionnaires (total duration is approximately 1 hour; administered at home; take place at baseline, 3, 6, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers can be spouses, relatives, or friends who care for and support the person with dementia without pay. If the caregiver does not live with the person with dementia, they have to visit the person with dementia at least 3 times a week to be eligible for the study.
* The person with dementia must be living at home cared for by the caregiver.
* The person with dementia should have a diagnosis of dementia or experience severe cognitive impairments suggesting dementia. Type of dementia is not an inclusion criterion.
* The person with dementia is not yet receiving formal care related to personal activities of daily living on account of his or her dementia more than once a week (defined by receiving assistance from a paid worker by e.g., health or social care professional as help with dressing/undressing; washing/bathing/showering; toileting; feeding/drinking; or taking medication).

Exclusion Criteria:

* Main exclusion criteria for both the caregiver and the person with dementia will be major mental or physical illness, such as major depression or stroke, that would affect their ability to participate in this study.
* Person with dementia or informal caregiver is participating in another intervention or similar support program.
* Dementia is caused by human immunodeficiency virus (HIV), acquired brain impairment, Down syndrome, chorea associated with Huntington's disease, or alcohol abuse.
* Inability to give informed consent will also be an exclusion criterion.
* Informal caregiver is younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Self-efficacy Scale (CSES) | 12 months
  The self-efficacy of informal caregivers measured by the Caregiver Self-efficacy Scale (CSES). This domain contains five items that are scored self-rated from 1 (not at all certain) to 10 (very certain) with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
TOPICS-MDS | 12 months
  Characteristics of the informal caregivers and persons with dementia collected by the TOPICS-MDS questionnaire to capture TOPICS-MDS:
  demographic characteristics, relation between informal caregiver and person with dementia, perseverance time (informal caregiver) instrumental and personal activities of daily living (person with dementia).
HADS | 12 months
  Depression and anxiety of informal caregivers measured by the Hospital and Anxiety Depression Scale (HADS). The HADS provides separate scores for depression and anxiety, each with 7 items on a four-point Likert scale ranging from 0 (not at all) to 3 (a great deal of the time). Total scores range from 0 to 21 per complaint, with higher scores indicating more anxiety or depression severity for the informal caregiver.
ICECAP-O | 12 months
  Quality of life of informal caregivers measured by the Investigating Choice Experiments for the Preferences of Older People CAPability measure for Older people (ICECAP-O). The ICECAP-O measures five capability attributes of quality of life: attachment, security, role, enjoyment, and control. All items are scored from 1 (no capability) to 4 (full capability), with higher scores indicating a higher overall quality of life for the informal caregiver.
QOL-AD | 12 months
  Quality of life of persons with dementia measured by the Quality of Life- Alzheimer's Disease scale (QOL-AD). The QOL-AD measures the quality of life for individuals with dementia on 13 separate items on a four-point Likert scale ranging from "poor" to "excellent" and was proxy-rated. Total scores range from 13 to 52 points, with higher total scores indicating a higher quality of life.
EDIZ | 12 months
  Experienced burden of informal caregivers measured by the EDIZ ("Ervaren Druk door Informele Zorg" / experienced burden of informal care). The EDIZ is a 9-item measurement for informal caregivers to assess self-perceived pressure from informal care. All items are scored on a five-point Likert scale ranging from 1 ("no!") to 5 ("yes!"), with higher scores indicating more perceived stress by the informal caregiver.
QDRS | 12 months
  Cognitive status of the person with dementia as estimated by the informal caregiver measured by a selection of the Quick Dementia Rating System (QDRS). The QDRS measures cognitive impairment for people with dementia and consists of six behavioral and four cognitive questions though, in this research, only the cognitive questions will be included proxy rated. These four items are scored on a scale from 0 to 3, with higher scores indicating more cognitive impairment.
EQ-5D-5L | 12 months
  Health-related quality of life of the informal caregiver (self-rated) and the person with dementia (proxy-rated) will be determined via the EQ-5D-5L assessment developed by EuroQol, which measures health-related quality of life on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a five-point Likert scale. The five responses provide a health profile indicated by a five-digit number, reflecting patient-reported categories across the dimensions. A higher score corresponds to more serious complaints, and thus a lower health-related quality of life for the informal caregiver.
RUD | 12 months
  Healthcare resource use of the informal caregivers and persons with dementia measured by the Resource Utilization in Dementia (RUD). This assessment measures the care resource use by the informal caregiver (self-rated) and the person with dementia (proxy-rated). For the caregiver, these resources include informal caregiver time (personal and instrumental activities of daily living and supervision), visits to care professionals, hospitalization, and productivity loss for those with a paid job. For the person with dementia, it covers accommodation (intermediate form, dementia-specific residential or long-term institutional care), visits to care professionals, hospitalizations, and social care services. The questions on medication usage were not included in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinische Neuropsychologie, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osstyn SL, Handels R, Boots LMM, Balvert SCE, Evers SMAA, de Vugt ME. The effectiveness and health-economic evaluation of "Partner in Balance," a blended self-management program for early-stage dementia caregivers: study protocol for a cluster-randomized controlled trial. Trials. 2023 Jun 22;24(1):427. doi: 10.1186/s13063-023-07423-9. PMID 37349828
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Fortinsky RH, Kercher K, Burant CJ. Measurement and correlates of family caregiver self-efficacy for managing dementia. Aging Ment Health. 2002 May;6(2):153-60. doi: 10.1080/13607860220126763. PMID 12028884
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Makai P, Looman W, Adang E, Melis R, Stolk E, Fabbricotti I. Cost-effectiveness of integrated care in frail elderly using the ICECAP-O and EQ-5D: does choice of instrument matter? Eur J Health Econ. 2015 May;16(4):437-50. doi: 10.1007/s10198-014-0583-7. Epub 2014 Apr 24. PMID 24760405
- [Background] Wimo A, Gustavsson A, Jonsson L, Winblad B, Hsu MA, Gannon B. Application of Resource Utilization in Dementia (RUD) instrument in a global setting. Alzheimers Dement. 2013 Jul;9(4):429-435.e17. doi: 10.1016/j.jalz.2012.06.008. Epub 2012 Nov 9. PMID 23142433
- [Background] Pot AM, van Dyck R, Deeg DJ. [Perceived stress caused by informal caregiving. Construction of a scale]. Tijdschr Gerontol Geriatr. 1995 Oct;26(5):214-9. Dutch. PMID 8750982